CLINICAL TRIAL: NCT04756908
Title: Evaluation of the Visual Performance and Safety of the Investigational Opira AIOL, A Commercial Multifocal IOL, and a Commercial Monofocal IOL
Brief Title: Safety and Effectiveness of the Opira AIOL in Comparison to Commercial IOLs in Patients Undergoing Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: FSV6, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIP-04
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opira AIOL (Experimental)
  Interventions: Device: Cataract Surgery
- Monofocal AIOL (Active Comparator)
  Interventions: Device: Cataract Surgery
- Multifocal AIOL (Active Comparator)
  Interventions: Device: Cataract Surgery

INTERVENTIONS:
Device: Cataract Surgery — The surgical procedure in which the natural crystalline lens is removed and replaced with a lens implant.

SUMMARY:
This is a clinical trial comparing an investigative accommodative IOL and two commercial IOLs in patients with cataracts undergoing primary cataract surgery.

DETAILED DESCRIPTION:
This is a prospective, multicenter clinical study comparing the safety and performance of the Opira accommodative IOL, a commercial monofocal IOL, and a commercial multifocal IOL. Eligible patients with bilateral cataracts will undergo cataract surgery implanting one of three study lenses, and will be followed postoperatively for 24 months

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 50-75 with bilateral cataracts, good potential vision, and clear intraocular media other than lens opacity

Exclusion Criteria:

* Comorbidities affecting visual acuity, IOP > 22mmHg, congential cataract

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 6 Months
Adverse event rates | 12 Months

CONTACTS AND LOCATIONS:
Locations (2):
- Clinica 2020, San José, Costa Rica
- Codet Vision Institute, Tijuana, Mexico